CLINICAL TRIAL: NCT01693341
Title: Caregiver-mediated Intervention in Home-living Chronic Stroke Patients
Brief Title: A Caregiver-mediated Intervention Improves the Functional Ability of Home-living Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CT-tsaiac1943
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Chronic stroke patients; Stroke rehabilitation; Caregiver; Caregiver-mediated intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care-giver mediated training (Active Comparator): Each patient and the caregiver of the intervention group received weekly home training and exercise counseling by a physical therapist about the caregiver mediated home exercise skill for stroke patient. The training program were progress weekly based on the patient's need.
  Interventions: Other: Care-giver mediated training
- Standard-care (No Intervention): Maintain the inherent standard-care

INTERVENTIONS:
Other: Care-giver mediated training — A physical therapist visited each subject and the caregiver (of the intervention group) once weekly for about 90 min/session to teach patient-skills and caregiver-skills. The therapist first reviewed the condition of each patient and planned patient-specific training programs, continuously performed 12 weeks.
  Arms: Care-giver mediated training

SUMMARY:
To examine the feasibility of improving stroke patients' physical functional recovery and social participation through improving caregiver's care capability.

DETAILED DESCRIPTION:
In the hospital, most rehabilitation units are like sheltered workshops and the therapists work with stroke patients in well-designed, but non-home-like, environment to improve the stroke patient's functional ability. After returning home, stroke patients face new challenges and also need to assume more responsibility for daily activities. Without continuing rehabilitation training or proper support, the patients can easily fall into a sedentary lifestyle and lead to declines in functional ability.However, providing home-based exercise by therapists directly would increase the health care cost and may not be practical for chronic stroke patients. Hence, the objective of the present study was to determine whether a caregiver-mediated, home-based intervention program is effective for improving stroke patients' functional ability and social participation.

ELIGIBILITY:
Inclusion Criteria:

1. >6 months post first stroke with mild to moderate disability (Brunnstrom stage III-V)
2. No longer undertaking active rehabilitation program(defined as ≤2 times/wk rehabilitation activities)

Exclusion Criteria:

1. Recurring strokes
2. Mental or cognitive impairment
3. Severe orthopedic disability or unstable medical conditions (such as severe rheumatoid arthritis or acute myocardial infarction)
4. Caregiver with mental/behavioral disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale | Baseline and 12 weeks
  Change from baseline in Stroke Impact Scale at 12 weeks

SECONDARY OUTCOMES:
10-meter walking speed | Baseline and 12 weeks
  Change from baseline in 10-meter walking speed (cm/sec) at 12 weeks
Berg balance scale | Baseline and 12 weeks
  Change from baseline in berg balance scale score at 12 weeks
6-min walking distance | Baseline and 12 weeks
  Change from baseline in 6-min walking distance at 12 weeks
Bathel index score | Baseline and 12 weeks
  Change from baseline in Bathel index score at 12 weeks
Lawton Instrumental Activities of Daily Living scale (IADL) | Baseline and 12 weeks
  Change from baseline in Lawton Instrumental Activities of Daily Living Scale at 12 weeks
Fugl-Meyer Assessment Scale | Baseline and 12 weeks
  Change frome baseline in Fugl-Meyer Assessment Scale score at 12 weeks

OTHER OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Baseline and 12 weeks
  Change from baseline in Center for Epidemiologic Studies Depression Scale score at 12 weeks
Caregiver Burden Scale | baseline and 12 weeks
  Change from baseline in Caregiver Burden Scale at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan. C Tsai, PhD, Study Chair — Asia University
Locations (1):
- St. Joseph Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Galvin R, Cusack T, O'Grady E, Murphy TB, Stokes E. Family-mediated exercise intervention (FAME): evaluation of a novel form of exercise delivery after stroke. Stroke. 2011 Mar;42(3):681-6. doi: 10.1161/STROKEAHA.110.594689. Epub 2011 Jan 13. PMID 21233462